CLINICAL TRIAL: NCT06055244
Title: Amantadine Therapy for Cognitive Impairment Related to Post-COVID Condition
Brief Title: Amantadine Therapy for Cognitive Impairment in Long COVID
Acronym: AmantadineLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Andrew Schamess, Associate Professor - Clinical, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023H0268; GF317855 (Other Grant/Funding Number: Private Donor)
Record Dates: First submitted 2023-09-22; First posted 2023-09-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Long COVID; Post-COVID19 Condition; Post-Acute COVID19 Syndrome
Keywords: long covid; PASC; post COVID condition; cognition; brain fog; amantadine
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue | interventions — Amantadine

STUDY DESIGN:
Intervention Model Description: Pilot randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amantadine (Experimental): Subjects will be treated with amantadine.
  Interventions: Drug: Amantadine
- Placebo (Placebo Comparator): Subjected received placebo identical to amantadine in appearance.
  Interventions: Drug: Amantadine

INTERVENTIONS:
Drug: Amantadine — Subjects will be give amantadine 100 mg twice daily.

SUMMARY:
This study will look at the effects of amantadine on cognitive function in persons with Long COVID. It will also collect specimens to study possible causes of cognitive symptoms in Long COVID, and whether any lab tests can predict who will respond better to amantadine.

DETAILED DESCRIPTION:
This study will enroll 60 subjects with Long COVID and cognitive symptoms such as problems with memory, concentration, speech and attention, and "brain fog." Subjects will be assigned randomly to two groups. One group will be treated with amantadine, the other group will receive placebo. The study will last 4 months. During that time, subjects will be assessed at regular intervals with symptom questionnaires, cognitive tests, and lab measurements.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and above at the signing of informed consent
2. Had a positive laboratory or home test for COVID19 within one year prior to signing of informed consent, with subsequent symptoms meeting criteria for PASC.
3. Subjective Cognitive impairment associated with PASC
4. Cognitive symptoms will be formally assessed at a pre-enrollment visit using the PROMIS Cognitive Function Questionnaire (CGQ) and the PROMIS Cognitive Abilities subset (CAS), which are validated patient-reported measures of subjective cognitive functioning. Potential participants must have a cumulative score less than 60 (indicating at least mild subjective cognitive dysfunction) to be eligible.
5. Is willing and able to comply with study visits and study-related procedures/assessments.
6. Is able to provide informed consent to participate in the study 5.
7. Is not currently taking a medication with adverse interactions with amantadine. (Table 2)
8. If the participant is of child bearing potential, , is not pregnant at enrollment based on negative urine pregnancy test.
9. If the participant is of child-bearing potential, is consistently using one or more forms of prescribed birth control, such as an oral contraceptive, intrauterine device or a long-acting reversible contraceptive.
10. Is not breastfeeding.
11. Is willing to abstain from alcohol use for the duration of the study.
12. Endorses self-reported cognitive impairment on the PROMIS CF[40].
13. Does not have any other contraindications to amantadine use as noted in section 6 below or as identified by the study clinician investigators.

Exclusion Criteria:

1. At risk for complications of study drug with conditions such as:

   * Lifetime history of compulsive or impulsive behavior: Compulsive gambling, hypersexuality, binge eating; suicidality.
   * Underweight, malnourished at time of enrollment.
   * History of restrictive eating disorder within 3 months prior to consent.
   * Lifetime history of heart failure or diagnosed cardiac arrhythmia.
   * Untreated angle closure glaucoma at time of enrollment.
   * Lifetime history of psychosis or psychotic disorder.
   * Lifetime history of seizure disorder.
   * Known allergy to amantadine.
   * History of binge drinking, heavy alcohol use, or alcohol use disorder as defined by the National Institute on Alcohol Abuse and Alcoholism (NIAAA)[54] and the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)[55].
   * Use of kava-kava within 3 months prior to consent.
   * Breastfeeding at screening or expected to be breastfeeding during study period.
   * Pregnant at time of screening or expecting to become pregnant during the study period.
2. Is taking a medication that adversely interacts with amantadine (see Table 2)
3. Has any physical examination findings, and/or history of any illness, concomitant medications or recent live vaccines that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the subject by their participation in the study.
4. Prior diagnosis of dementia, neurodegenerative disorder, multiple sclerosis or other autoimmune neurologic disorder, or cognitive impairment.
5. Enrolled in any other research study involving intervention for PASC.
6. If the individual is of child-bearing potential, is not consistently using one or more forms of prescribed birth control.
7. Is not willing to abstain from alcohol for the duration of the study.
8. Is not willing and able to adhere to study visits and study-related procedures/assessments.
9. Is not able to provide informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Improvement in cognitive symptoms | 4 months
  Improvement in scores on self-assessment of overall cognitive functioning
Improvement on objective cognitive testing | 4 months
  Subjects will be administered battery of cognitive tests to determine if there is a change in objective cognitive function

SECONDARY OUTCOMES:
Mood symptoms | 4 months
  Subjects will be administered anxiety and depression questionnaires to determine if there is improvement in mood symptoms.
Medication tolerability | 4 months
  Subjects will complete a questionnaire addressing tolerability of amantadine and side effects experienced

CONTACTS AND LOCATIONS:
Overall Officials: Andrew I Schamess, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there will be a plan to make IPD available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon study completion
Access Criteria: As appropriate